CLINICAL TRIAL: NCT02473341
Title: Gut-Liver Axis Modulation With IgG-Enriched Immunotherapy in Severe Alcohol-Associated Hepatitis: A Multicentre, Randomised, Placebo-Controlled Trial
Brief Title: Gut-Liver Axis Modulation With IgG-Enriched Immunotherapy in Severe Alcohol-Associated Hepatitis
Acronym: BC-SAAH
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dayanand Medical College and Hospital (Other)
Responsible Party: Principal Investigator, Prof. Sandeep S Sidhu, Prof. Sandeep Singh Sidhu, Dayanand Medical College and Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMCH/R&D/2017/578
Record Dates: First submitted 2015-06-08; First posted 2015-06-16 (Estimated); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Alcoholic Hepatitis
Keywords: Bovine Colostrum; Endotoxin; MELD; mDF; Alpha TNF
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bovine colostrum (Experimental): Protein 1.5 gm/kg/day, energy (kcal) 30-40/day, B complex vitamins daily. Pasteurized Bovine colostrum as a lyophilised freeze dried powder (20 gm thrice a day) for 4 weeks.
  + Antibiotics + Diuretics +Terlipressin for HRS + acid suppression for prophylaxis against gastrointestinal hemorrhage + EVL for variceal bleed +drugs for HE if indicated
  Interventions: Drug: Bovine Colostrum
- Placebo (Placebo Comparator): Placebo (Pasteurised Milk Powder) 20 gms thrice a day for 4 weeks Protein 1.5 gm/kg/day, energy (kcal) 30-40/day, B complex vitamins daily.
  + Antibiotics + Diuretics + drugs for HE + Terlipressin for HRS + acid suppression for prophylaxis against gastrointestinal hemorrhage + EVL for variceal bleed + if indicated.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bovine Colostrum — Protein 1.5 gm/kg/day, energy (kcal) 30-40/day, B complex vitamins daily. Pasteurized Bovine colostrum as a freeze dried powder (20 gm thrice a day) for 4 weeks.
  + Antibiotics + Diuretics +Terlipressin for HRS + acid suppression for prophylaxis against gastrointestinal hemorrhage + EVL for variceal bleed +drugs for HE if indicated
  Arms: Bovine colostrum
Drug: Placebo — Protein 1.5 gm/kg/day, energy (kcal) 30-40/day, B complex vitamins daily. Placebo (Pasteurised Milk Powder) 20 gms thrice a day for 4 weeks
  + Antibiotics + Diuretics + drugs for HE + Terlipressin for HRS + acid suppression for prophylaxis against gastrointestinal hemorrhage + EVL for variceal bleed + if indicated.
  Arms: Placebo

SUMMARY:
Severe alcohol-associated hepatitis is associated with hepatocellular necrosis, inflammation, hyperactivated immune system, paradoxical immune exhaustion, leaky gut, and alteration in the gut microbiome. The leading cause of mortality is a bacterial infection with multi-organ failure.

Pentoxifylline was ineffective and Interleukin-1-based therapies - Anakinra and Canakinumab have not improved survival rates. The granulocyte colony-stimulating factor has shown mixed results. Indian studies improved 90-day survival, while Western studies on Pegfilgrastim have been negative. Corticosteroids decrease the mortality for only a month. In a recent study on Severe alcohol-associated hepatitis, Larsucosterol, a DNA methyltransferase inhibitor, was associated with non-significant improvement in 90-day mortality: 14.7 % (30 mg/day) and 16.67 % (90 mg/day) versus 24.27% on Methylprednisolone. Thus, a more durable treatment of severe alcohol-associated hepatitis is needed.

Bovine Colostrum contains many bioactive components such as immunoglobulin G, A, and M (70 - 80 % of total protein), Lactoferrin and Short-chain fatty acids. Bovine Colostrum has 30-100 times higher Lactoferrin concentration than milk. IgG and Lactoferrin synergistically neutralise lipopolysaccharide/ Endotoxin and act on mucosa-associated lymphoid tissue of the leaky gut, transforming it into healthy mucosa.

Fewer bacteria and Endotoxins - Pathogen-associated molecular patterns enter the portal circulation to interact with Toll-Like Receptor - 4 of the Liver Kupffer cells. Proinflammatory cytokines such as interleukins-1,6,8 and tumour necrosis factor-alpha, generation decreases, mitigating hepatocyte inflammation, necrosis, and cell death. In this study, we aimed to assess the effectiveness and safety of Gut-Liver Axis Modulation with IgG-Enriched Oral Immunotherapy(Bovine Colostrum) in Severe Alcohol-Associated Hepatitis

DETAILED DESCRIPTION:
INTRODUCTION

Background and Rationale Severe alcoholic hepatitis (AH) imposes a significant global burden, markedly contributing to liver-related illness and death. The worldwide impact is driven by increasing alcohol consumption and the lack of effective treatments for severe cases. Chronic alcohol intake disrupts normal gut microbiome balance, leading to dysbiosis. This imbalance involves an increase in harmful bacteria and a decrease in beneficial ones, affecting overall gut health. Alcohol also damages the intestinal barrier, making it more permeable. This increased permeability allows bacteria and their harmful byproducts, such as lipopolysaccharides (LPS), to leak into the bloodstream. The leaked bacteria and LPS (pathogen-associated molecular patterns-PAMPs) reach the liver via the portal vein. In the liver, LPS activates toll-like receptor 4 (TLR4) on immune cells, triggering a pro-inflammatory response and hepatocyte necrosis. These PAMPs also contribute to systemic endotoxemia and septicaemia. Despite optimal medical therapy, often including prednisolone, severe alcohol-associated hepatitis has a 28-day mortality rate of 30-40%. The gut-liver axis has emerged as a promising target for treatment in sAH. Interventions such as antibiotics, nonabsorbable disaccharides, probiotics, and fecal microbiota transplantation have shown variable benefits in modulating intestinal permeability and microbial imbalance in cirrhosis. However, none are currently standard treatments for sAH. Furthermore, corticosteroids, while somewhat improving short-term survival, do not address the gut-driven inflammatory cascade and may increase the risk of infections. Bovine colostrum, the first milk produced after birth, is naturally rich in immunoglobulin G (IgG), lactoferrin, antimicrobial peptides, and short-chain fatty acids. Preclinical studies show that oral bovine colostrum can neutralize lipopolysaccharides, promote epithelial regeneration transforming the leaky gut into a healthy mucosal barrier, and modify the intestinal microbiota. These properties are highly relevant to reducing the pathogenic factors of sAH. Therefore, we conducted a multicenter, double-blind, placebo-controlled Phase 3 trial to determine whether adding oral IgG-enriched bovine colostrum to standard medical treatment could enhance survival and liver function in patients with sAH. Our hypothesis was that targeting the gut-liver axis with a safe, enterally delivered biologic would decrease systemic and hepatic inflammation, mitigate hepatocyte necrosis, lower infection rates, and improve clinical outcomes.

Natural History of Severe Alcohol-Associated Hepatitis in the West:

In the STOPAH study, 60% - 67% patients were males; baseline Maddrey's Discriminant Function was 61.9 + 25.7 and the Model For End-Stage Liver Disease was 20.7 + 5.5 in the Placebo arm. Out of the total 418 deaths, 168(40%) occurred before day 29, 28% occurred between days 28 and 90 , 32% occurred between day 91 and 1 year.

Background cirrhosis was in 86.2-93.7% patients with Severe Alcohol Associated Hepatitis treated with prednisone who had undergone liver biopsies

Natural History of Severe Alcohol-Associated Hepatitis in India:

In all Indian studies patients had a very severe disease as evidenced by the high Maddrey's Discriminant Function scores and Model For End-Stage Liver Disease scores. The majority of deaths occurred within the first month, with only a few deaths in the second and third months. The vast majority of these patients had underlying cirrhosis and were males. Corticosteroids could be offered in only 12%, due to contraindications in the rest of the patients - Acute Kidney Injury (37%) , infection (45%), Gastrointestinal bleed in (18%), patient's refusal in 17%.

Treatment Abstinence from alcohol This is the most important factor in predicting the outcome after surviving the acute Alcohol-Associated hepatitis (AH) episode.

Nutrition A careful evaluation of nutritional status and energy intake is done, with the aim to deliver 35-40 kcal/kg of body weight and a daily protein intake of 1.2-1.5 g/kg of body weight orally. Small frequent meals and a bedtime snack is advised. Supplementation of Thiamine, other B vitamins, Vitamin D, and trace elements, including Zinc, should be done.

Pharmacotherapy of Severe Alcohol-Associated Hepatitis Corticosteroids All recent Western studies have concluded that corticosteroid use decreases the 30-day, but not 90- or 180-day mortality rate in patients with Severe Alcohol-Associated Hepatitis. A more durable treatment of severe alcohol-associated hepatitis is needed. The Maddrey's Discriminant Function in the Western studies ranged from [Median (Inter Quartile Range)] 54.4 (39.2 - 76.1) to 69.7(53.7 - 89.4). The Model For End-Stage Liver Disease score ranged from [median (Inter Quartile Range)] 21.49 (19.95 - 22.89) to 25(22 - 27). The 90- day mortality rate was 30% in the STOPAH trial, 30% in the DASH trial and 26% in the AntiBiocor trial compared to 10% in the Gawrieh S, et al study due to younger patients in the last study. The pooled 90-day survival was 73.61% (95% CI: 68.18%-78.69%) in placebo-treated patients in above studies.

Combining four contemporary Indian studies on Severe Alcohol-Associated Hepatitis, the median Maddrey's Discriminant Function scores ranged from 70 (32 - 320) to 84 (56 - 185) and the median Model For End-Stage Liver Disease scores ranged from 26 (15 - 40) to 27.5 (19 - 41). The 90-day survival ranged from 22% - 56% on standard medical treatment.

The inference is that Severe Alcohol-Associated Hepatitis in Indian patients is more severe than in Western patients.

Hence, in light of the National Institute on Alcohol Abuse and Alcoholism recommendations, it is clear that Corticosteroids are not a therapeutic option for Indian patients as Maddrey's Discriminant Function and Model For End-Stage Liver Disease scores are very high.

Although our pilot study conducted in 2015 had shown that treatment with a combination of Bovine Colostrum and Corticosteroids had improved the Maddrey's Discriminant Function level and survival rate at 3 months significantly, we would only use Bovine Colostrum as a therapeutic option versus standard medical treatment, rather than use corticosteroids as a active comparator arm which has no impact on the 90-day mortality.

Larsucosterol Larsucosterol, an endogenous oxysterol, is an epigenetic inhibitor of DNA methyltransferases, mitigating apoptosis. In a recent study (Model of End-Stage Liver Disease score-24, Maddrey's discriminant function scores 57.2 - 63), Larsucosterol was associated with non-significant improvement in 90-day mortality: 15.2 % (30 mg/day) and 16.8 % (90 mg/day) versus 24.5% on Methylprednisolone. However, the severity of hepatitis was milder compared to Indian our studies.

Failed Treatments Pentoxifylline was ineffective, and Interleukin-1-based therapies - Anakinra and Canakinumab have not improved survival rates. The granulocyte colony-stimulating factor has shown mixed results. Indian studies improved 90-day survival, while Western studies on Pegfilgrastim have been negative.

Bovine colostrum Composition and Rationale for its Treatment Potential in Severe Alcohol-Associated Hepatitis The Bovine Colostrum has the following components: fat, protein, peptides, lactose ,immunoglobins, lactoferrin, lysozyme, lactoperoxidase, insulin growth factor-I .

Colostrum contains elevated levels of IgG, IgA, and IgM, which make up 70-80% of the total protein in colostrum. Short-Chain Fatty Acids in Colostrum improve the integrity of the intestinal inner cell membrane. The lactoferrin concentration in colostrum is 30 - 100 fold higher than that in milk.

Lactoferrin binds to lipid A of Lipopolysaccharide (LPS) to neutralize it. IgG and lactoferrin synergistically neutralize LPS. IgG and lactoferrin interact with mucosa-associated lymphoid tissue of leaky mucosal barrier to convert into healthy mucosal barrier. It increases the growth and proliferation of enterocytes.

Additionally, lactoferrin has an impact on the levels of cytokines and chemokines that are produced by Gut-Associated Lymphoid Tissue and creates an environment for the growth of beneficial bacteria in the gut. Fewer bacteria and LPS /Endotoxin, - pathogen-associated molecular particles enter the Portal vein resulting in decreased trafficking and interaction of bacteria and LPS with Toll-like receptors-4 of the macrophages and Kupffer Cells in the liver. The production of pro-inflammatory cytokines such as interleukin-1 beta,6,8,10, (IL-1 beta,6,8,10), Reactive Oxygen Species (ROS) and Tumour necrosis factor-alpha (TNF-alpha) are decreased and hepatocellular necrosis is mitigated.

Thermal processing of colostrum In studies conducted by Donahue and Godden et al., heating colostrum at 60 °C for 60 min decreased total plate counts, coliform counts and other pathogens, but did not affect native IgG concentration.

Derivation of Dose of Bovine Colostrum Oral bovine colostrum preparation (Lactobin®) 56g/day was given prophylactically to 20 patients for 3 days preoperatively who underwent abdominal surgeries, and (Placebo) standard milk 56 g/day was given for 3 days to 20 similar patients.

The course of the plasma endotoxin / LPS levels and the endotoxin neutralization capacity were measured daily up to the 10th postoperative day. The results showed that the LPS levels in the Lactobin group, were significantly lower than those in the control group (p < 0.05). The difference between the two groups was apparent on the day of the operation and the day after. There was a significantly greater increase in endotoxin-neutralizing capacity in the patients treated with lactobin than in the control group (p<0.006). Thus, Bovine Colostrum has been successfully used to decrease the level of Endotoxemia / Lipopolysaccharides.

In the second placebo-controlled randomized study, 60 patients who underwent coronary bypass operations with either 42 g of a Bovine colostrum milk preparation per day or placebo for 2 days preoperatively. There was no reduction in Endotoxin levels and no increase in endotoxin-neutralizing capacity levels in patients receiving the lower dose of Colostrum. Thus, the correct dose of Bovine Colostrum appears to be 60 grams/day.

The protein content of the Bovine Colostrum used in our study was 52.75% and the IgG content was 34.25% (342.5 mg IgG/gram) of protein The protein content was 80% and the IgG/gram of the total Protein content was 52 mg in Lactobin® Bovine Colostrum. Thus, the Colostrum used in our study has a much higher content of IgG than the Lactobin Colostrum used by Bolke E et al. This is because the Spray dried technique used in Lactobin preparation decreases the IgG much more than the freeze-dried technique used in the preparation of Bovine Colostrum in the current study.

Trial design This is a multicentre, parallel, double-blind, randomised (1:1), placebo-controlled trial.

Methods: Participants Study setting The study will recruit patients admitted with "probable" Severe Alcohol-Associated Hepatitis at five academic centers and Hospitals in India. The accuracy of a clinical diagnosis of "probable Alcohol-Associated Hepatitis using the Crabbe et al criteria is 96%. Thus patients can be started on initiating treatment promptly on presentation rather than to rely upon histology which may delay assessment .Hence , no patients underwent liver biopsy.

Relevant concomitant care given during the trial Standard of care treatment will be given in both arms are as follows- Oral / Enteral nutrition (if oral intake is insufficient: Protein 1.2 -1.5 gm/kg/day, energy (kcal) 35-40/day, small frequent feeds with a bedtime snack of 50 g of complex carbohydrates with 13.5 g of proteins and B complex vitamins daily. Antibiotics for sepsis; Salt restriction and Diuretics for Ascites; Lactulose / Rifaximin / L Ornithine L Aspartate for Hepatic Encephalopathy; Terlipressin and Albumin for Type 1 Hepato Renal Syndrome; Carvedilol for prophylaxis against variceal hemorrhage; Terlipressin with Endoscopic Variceal Ligation for variceal bleed, if indicated.

Criteria for discontinuing or modifying allocated interventions for a given trial participant Occurrence of adverse effects of Bovine colostrum (Experimental arm) and pasteurised milk powder (placebo comparator): Allergy, Lactose Intolerance Strategies to improve adherence to intervention protocols All patients will be initially admitted to the hospital ICU / wards. After discharge from the hospital, the patients will be contacted telephonically and reminded to shall return for outpatient visits after 7 days, 14 days, 21 days, 28 days, and then bimonthly for two months. At the outpatient visit, history, physical examination, and laboratory tests will be done. The patients will return the empty sachets (which will be counted), and a new batch of sachets will be given until the next outpatient visit

Investigations

Each patient shall have an:

1. Abdominal ultrasonography.
2. Laboratory tests: Hemogram, prothrombin time, Procalcitonin levels, blood glucose, liver function tests, blood urea, serum creatinine, and serum electrolytes will be done at baseline, and at 7 days, 14 days, 21 days, 28 days, and then bimonthly for two months or earlier, if indicated.
3. Microbiologic tests: Blood, urine, sputum cultures, and cultures of aspirates from endotracheal tubes in ventilated patients shall be performed at admission. At baseline, a diagnostic paracentesis will be performed in all patients with ascites
4. Cytokine levels: Endotoxin, Tumor Necrosis Factor-alpha, Interleukin 6 & 8 levels will be done at baseline and end of treatment
5. Tests of Aetiology : To rule out viral, autoimmune hepatitis, Wilson disease, Hemochromatosis and Non-alcoholic steatohepatitis will be done.

i. Assessment of effect of Intervention on Intestinal Barrier function: Serum Endotoxin levels as well as the TNF -alpha levels (an important downstream pro-inflammatory mediator).

Sample size determination In an Indian study of patients suffering from Severe Alcohol-Associated Hepatitis, published in 2014 by Singh et al the the Maddrey Discriminant Function score was 77.4 (range: 37- 235), the Model for End-Stage Liver Disease score was 27.5 (range:19- 41), and the survival rate was 22% at 90 days.

Hence, in our study of patients with Severe Alcohol-Associated Hepatitis, we calculated the sample size based on the above study.

We considered a 20% increase in survival rate (80% power at 5% alpha), to be clinically meaningful and sufficient to change practice. To detect a 20% increase in survival (from 22% to 42%) in 3 months [the sample size was based on survival at a fixed time point (22% vs 42% at 3 months)], we required 79 patients in each group. Assuming, 10% dropouts. the total sample size required for the study is 174.

Randomisation Consecutive patients diagnosed with Severe Alcohol-Associated hepatitis will be then registered by the site medical team onto the trial site via Trans European Network for clinical trials services, a web-based registration and randomisation system, and randomised into two groups (groups A and B) to receive active drug or placebo 1:1.

Blinding Treatment allocation will be blinded to patients, investigators, data collectors, and statisticians by providing each patient with a unique number from the Trans European Network for clinical trials services registration system

Statistical methods Statistical methods for primary and secondary outcomes

Subject population (S) for analysis:

For primary survival (efficacy) analysis, we will use intention-to-treat analysis, in such a way that all study subjects who are randomized, regardless of adherence to study medication, will be used in the analysis in the treatment arms to which they are originally assigned to at randomization ("as randomized"). Significance will be assessed using a two-sided alpha level of 0.05.

Baseline Patients' Characteristics The baseline patients' characteristics will be compared between the two treatment groups to demonstrate the actual study group balance and to ensure whether a proper randomization is established or not. We will measure central tendency and variability with means and standard deviations or medians and interquartile range for continuous characteristics and frequencies with percentages for categorical characteristics.

Primary Outcome Unadjusted Log-Rank Test Of The Kaplan-Meier Survival Estimates This test for the two treatment arms has a at a two-sided alpha level of 0.05 with survival censored at 3 months.

Hazard Ratios Further, a Cox proportional hazards regression model (with survival censored at 3 months) will be used to estimate the hazard ratio with a 95% confidence interval associated with the treatment arm (A) compared to the Placebo (B).

Scaled Schoenfeld Residuals plots The pattern against the time in these plots will be observed. If a nonrandom pattern is observed, this will be considered a violation of the Proportional Hazards assumption.

Restricted Mean Survival Time To address the violation of the proportional hazards assumption, the restricted mean survival time for both treatment arms over 90 days for the Actual Observed outcome and the Worst Case Scenario will be calculated.

Secondary Outcomes A similar unadjusted log-rank test of the Kaplan-Meier survival estimates and Cox proportional hazards regression model analysis will be planned for secondary outcome survival at 1 month. In the graphical Scaled Schoenfeld tests, the pattern against the time in these plots will be observed. If a non-random pattern is observed ,we will then calculate the restricted mean survival time for both treatment arms over 30 days for the Actual Observed outcome and the Worst Case Scenario.

Other secondary outcomes measures such as Change in Maddrey Discriminant Factor levels/ Model For End-Stage Liver Disease score, Endotoxin levels, and Cytokines levels between baseline and 4 weeks assessment will be assessed for normal distribution by graphical (Quantile-Quantile Plot) interpretation and numerical method (Kolmogorov-Smirnov test). A paired t-test will be used for all those outcomes which will follow approximately normal distribution and a Mann-Whitney U test will be used for skewed parameters. The proportionality assumption will be assessed for the considered ordinal outcome number of episodes of sepsis (Pneumonia, Spontaneous Bacterial Peritonitis, cellulitis, and Urinary Tract Infection, Bacteremia). Partial proportional odds ratio regression will be used to assess the effect of treatment on the number of episodes of sepsis (Pneumonia, Spontaneous Bacterial Peritonitis, Cellulitis, Urinary Tract Infection, Bacteremia) over 4 weeks.

Subgroup analysis Subgroup analysis may be conducted based on the clinical age group , grams of alcohol consumed criteria, alcohol relapse (recidivism) and the Model for End-Stage Liver Disease scores.

Sensitivity Analysis Sensitivity analyses will be performed to assess the robustness of the results to protocol deviations.

Unadjusted and Adjusted (For Centre, Acute Kidney Injury, and Ascites grade) Relative Risk of mortality- will be performed for :

* Actual Observed Outcomes
* Best-case scenario assumption - participants lost to follow-up are considered alive in the Colostrum arm and deceased in the Placebo group
* Worst-case scenario assumption - participants lost to follow-up are considered deceased in the Colostrum arm and alive in the Placebo group.

Interim analyses No formal interim analysis is planned for this trial. Monitoring for Adverse Events A treatment-emergent Adverse Event will be defined as an Adverse Event that begins or that worsens in severity after at least one dose of the study drug has been administered. Any adverse event occurring during the study will be documented in the subject's Case Report Form specifying the time of onset, the duration, the severity, and the relationship to the test medication

Grades of Severity of the Adverse Event as per the Common Terminology Criteria for Adverse Events (CTCAE) v 5.0:

* Grade 1 Mild Adverse Event
* Grade 2 Moderate Adverse Event
* Grade 3 Severe Adverse Event
* Grade 4 Life-threatening or disabling Adverse Event
* Grade 5 Death related to Adverse Event.

ELIGIBILITY:
Inclusion Criteria:

* Onset of jaundice within prior 8 weeks
* Ongoing consumption of > 40 (female) or 60 (males) g alcohol/day for 6 months or more, with less than 60 days of abstinence before the onset of jaundice
* Aspartate aminotransferase > 50, aspartate aminotransferase/alanine aminotransferase > 1.5, and both values < 400 IU/L
* Serum bilirubin (total) > 3.0 mg/dL
* Liver biopsy confirmation in patients with confounding factors including possible ischemic hepatitis (eg, severe upper gastrointestinal bleed, hypotension, or cocaine use within 7 days); possible DILI; uncertain alcohol use assessment (eg, patient denies excessive alcohol use); and atypical laboratory tests (eg, AST < 50 IU/mL or > 400 IU/mL, AST/ALT ratio < 1.5), antinuclear antibody > 1:160 or SMA > 1:80
* Maddrey's discriminant function ≥ 32 assuming a control prothrombin time of 12 seconds
* Model for End-stage Liver Disease score > 20

Exclusion Criteria

* Uncontrolled infections
* Multiorgan failure
* Uncontrolled upper gastrointestinal bleeding. "However, patients with recent Upper Gastro Intestinal bleeding, without significant hypotension that is controlled for >48 hours, will be included in the study."
* Preexisting kidney injury with serum creatinine > 2.5 mg/dL
* Other underlying liver diseases including hepatitis B infection,* autoimmune liver diseases, Wilson disease, suspected drug-induced liver injury*
* Hepatocellular carcinoma or other active malignancies except skin cancer
* Pregnancy
* Uncontrolled drug addiction
* Cow milk allergy or severe lactose intol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 3 month
  Survival at 3 month

SECONDARY OUTCOMES:
Change in mDF and MELD levels | one month
  Change in mDF and MELD levels will be measured at baseline and after 30 days of treatment
Change in Endotoxin levels | one month
  Change in Endotoxin levels will be measured at baseline and after 4 weeks of treatment
Change in Cytokines levels | one month
  Change in Cytokines levels will be measured at baseline and after 30 days of treatment
Number of episodes of sepsis | 1 month
  Number of episodes of sepsis (bacteremia, Pneumonia, SBP, Cellulitis, UTI) [Criteria for defining infections in cirrhosis are appropriate for Severe Alcohol-Associated Hepatitis] {32. Bajaj JS, O'Leary JG, Reddy KR, Wong F, Olson JC, Subramanian RM, Brown G, Noble NA, Thacker LR, Kamath PS; NACSELD. Second infections independently increase mortality in hospitalized patients with cirrhosis: the North American consortium for the study of end-stage liver disease (NACSELD) experience. Hepatology. 2012 Dec;56(6):2328-35. doi: 10.1002/hep.25947. PMID: 22806618; PMCID: PMC3492528.}
Survival | 1 month
  Survival at 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Singh Sidhu, DM, Principal Investigator — Dayanand Medical College and Hospital, Ludhiana, Punjab, India; Ajay Duseja, DM, Principal Investigator — PGI Hospital, Chandigarh, India; Shalimar S, DM, Principal Investigator — All India Institute of Medical Sciences; Dharmesh Kapoor, Principal Investigator — Gleneagles Global Hospital, Hyderabad; Sandeep Nijhawan, Principal Investigator — SMS Hospital, Jaipur, India
Locations (5):
- India (5):
  - Department of Gastroenterology, Dayanand Medical College and Hospital, Ludhiana, Punjab
  - Post Graduate Medical Institute of Medical Education and Research, Chandigarh
  - Department of Hepatology, Global Hospital, Hyderabad
  - Sawai Man Singh Medical College, Jaipur
  - All India Institute of Medical Sciences, New Delhi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Feng D, Hwang S, Guillot A, Wang Y, Guan Y, Chen C, Maccioni L, Gao B. Inflammation in Alcohol-Associated Hepatitis: Pathogenesis and Therapeutic Targets. Cell Mol Gastroenterol Hepatol. 2024;18(3):101352. doi: 10.1016/j.jcmgh.2024.04.009. Epub 2024 May 1. PMID 38697358
- [Background] Karakike E, Moreno C, Gustot T. Infections in severe alcoholic hepatitis. Ann Gastroenterol. 2017;30(2):152-160. doi: 10.20524/aog.2016.0101. Epub 2016 Oct 27. PMID 28243035
- [Background] Thursz MR, Richardson P, Allison M, Austin A, Bowers M, Day CP, Downs N, Gleeson D, MacGilchrist A, Grant A, Hood S, Masson S, McCune A, Mellor J, O'Grady J, Patch D, Ratcliffe I, Roderick P, Stanton L, Vergis N, Wright M, Ryder S, Forrest EH; STOPAH Trial. Prednisolone or pentoxifylline for alcoholic hepatitis. N Engl J Med. 2015 Apr 23;372(17):1619-28. doi: 10.1056/NEJMoa1412278. PMID 25901427
- [Background] Louvet A, Thursz MR, Kim DJ, Labreuche J, Atkinson SR, Sidhu SS, O'Grady JG, Akriviadis E, Sinakos E, Carithers RL Jr, Ramond MJ, Maddrey WC, Morgan TR, Duhamel A, Mathurin P. Corticosteroids Reduce Risk of Death Within 28 Days for Patients With Severe Alcoholic Hepatitis, Compared With Pentoxifylline or Placebo-a Meta-analysis of Individual Data From Controlled Trials. Gastroenterology. 2018 Aug;155(2):458-468.e8. doi: 10.1053/j.gastro.2018.05.011. Epub 2018 May 5. PMID 29738698
- [Background] Szabo G, Mitchell M, McClain CJ, Dasarathy S, Barton B, McCullough AJ, Nagy LE, Kroll-Desrosiers A, Tornai D, Min HA, Radaeva S, Holbein MEB, Casey L, Cuthbert J. IL-1 receptor antagonist plus pentoxifylline and zinc for severe alcohol-associated hepatitis. Hepatology. 2022 Oct;76(4):1058-1068. doi: 10.1002/hep.32478. Epub 2022 Jun 2. PMID 35340032
- [Background] Gawrieh S, Dasarathy S, Tu W, Kamath PS, Chalasani NP, McClain CJ, Bataller R, Szabo G, Tang Q, Radaeva S, Barton B, Nagy LE, Shah VH, Sanyal AJ, Mitchell MC; AlcHepNet Investigators. Randomized trial of anakinra plus zinc vs. prednisone for severe alcohol-associated hepatitis. J Hepatol. 2024 May;80(5):684-693. doi: 10.1016/j.jhep.2024.01.031. Epub 2024 Feb 10. PMID 38342441
- [Background] Vergis N, Patel V, Bogdanowicz K, Czyzewska-Khan J, Keshinro R, Fiorentino F, Day E, Middleton P, Atkinson S, Tranah T, Cross M, Babalis D, Foster N, Lord E, Quaglia A, Lloyd J, Goldin R, Rosenberg W, Parker R, Richardson P, Masson S, Whitehouse G, Sieberhagan C, Patch D, Naoumov N, Dhanda A, Forrest E, Thursz M. IL-1 Signal Inhibition in Alcohol-Related Hepatitis: A Randomized, Double-Blind, Placebo-Controlled Trial of Canakinumab. Clin Gastroenterol Hepatol. 2025 Apr;23(5):797-807.e5. doi: 10.1016/j.cgh.2024.07.025. Epub 2024 Aug 23. PMID 39181422
- [Background] Singh V, Sharma AK, Narasimhan RL, Bhalla A, Sharma N, Sharma R. Granulocyte colony-stimulating factor in severe alcoholic hepatitis: a randomized pilot study. Am J Gastroenterol. 2014 Sep;109(9):1417-23. doi: 10.1038/ajg.2014.154. Epub 2014 Jun 17. PMID 24935272
- [Background] Singh V, Keisham A, Bhalla A, Sharma N, Agarwal R, Sharma R, Singh A. Efficacy of Granulocyte Colony-Stimulating Factor and N-Acetylcysteine Therapies in Patients With Severe Alcoholic Hepatitis. Clin Gastroenterol Hepatol. 2018 Oct;16(10):1650-1656.e2. doi: 10.1016/j.cgh.2018.01.040. Epub 2018 Jan 31. PMID 29391265
- [Background] Shasthry SM, Sharma MK, Shasthry V, Pande A, Sarin SK. Efficacy of Granulocyte Colony-stimulating Factor in the Management of Steroid-Nonresponsive Severe Alcoholic Hepatitis: A Double-Blind Randomized Controlled Trial. Hepatology. 2019 Sep;70(3):802-811. doi: 10.1002/hep.30516. Epub 2019 Mar 25. PMID 30664267
- [Background] Tayek JA, Stolz AA, Nguyen DV, Fleischman MW, Donovan JA, Alcorn JM, Chao DC, Asghar A, Morgan TR; Southern California Alcoholic Hepatitis (SCAH) Consortium. A phase II, multicenter, open-label, randomized trial of pegfilgrastim for patients with alcohol-associated hepatitis. EClinicalMedicine. 2022 Oct 12;54:101689. doi: 10.1016/j.eclinm.2022.101689. eCollection 2022 Dec. PMID 36267499
- [Background] Sidhu SS, Goyal O, Singla P, Gupta D, Sood A, Chhina RS, Soni RK. Corticosteroid plus pentoxifylline is not better than corticosteroid alone for improving survival in severe alcoholic hepatitis (COPE trial). Dig Dis Sci. 2012 Jun;57(6):1664-71. doi: 10.1007/s10620-012-2097-4. Epub 2012 Mar 3. PMID 22388710
- [Background] Louvet A, Labreuche J, Dao T, Thevenot T, Oberti F, Bureau C, Paupard T, Nguyen-Khac E, Minello A, Bernard-Chabert B, Anty R, Wartel F, Carbonell N, Pageaux GP, Hilleret MN, Moirand R, Nahon P, Potey C, Duhamel A, Mathurin P. Effect of Prophylactic Antibiotics on Mortality in Severe Alcohol-Related Hepatitis: A Randomized Clinical Trial. JAMA. 2023 May 9;329(18):1558-1566. doi: 10.1001/jama.2023.4902. PMID 37159035
- [Background] Pavlov CS, Varganova DL, Casazza G, Tsochatzis E, Nikolova D, Gluud C. Glucocorticosteroids for people with alcoholic hepatitis. Cochrane Database Syst Rev. 2019 Apr 9;4(4):CD001511. doi: 10.1002/14651858.CD001511.pub4. PMID 30964545
- [Background] Shiffman M, Da B, Goel A, Kwong A, Stein L, Moreno C, Nicoll A, Mehta A, Louvet A, Flamm S, Pyrsopoulos N, Satapathy S, Kuo A, Ganger D, Aloman C, Strasser SI, Tse E, Russo MW, Rockey D, Gray M, Mitchell M, Thursz M, Krebs W, Scott D, Blevins C, Ellis D, Brown J, Sussman N, Lin W. Larsucosterol for the Treatment of Alcohol-Associated Hepatitis. NEJM Evid. 2025 Feb;4(2):EVIDoa2400243. doi: 10.1056/EVIDoa2400243. Epub 2025 Jan 28. PMID 39873544
- [Background] Thursz M, Mathurin P. Targeting IL-1 in severe alcohol-related hepatitis: How many frogs will we need to kiss to find an effective therapy? J Hepatol. 2024 May;80(5):678-680. doi: 10.1016/j.jhep.2024.03.011. Epub 2024 Mar 16. No abstract available. PMID 38499249
- [Background] Struff WG, Sprotte G. Bovine colostrum as a biologic in clinical medicine: a review--Part II: clinical studies. Int J Clin Pharmacol Ther. 2008 May;46(5):211-25. doi: 10.5414/cpp46211. PMID 18538107
- [Background] Liu N, Feng G, Zhang X, Hu Q, Sun S, Sun J, Sun Y, Wang R, Zhang Y, Wang P, Li Y. The Functional Role of Lactoferrin in Intestine Mucosal Immune System and Inflammatory Bowel Disease. Front Nutr. 2021 Nov 25;8:759507. doi: 10.3389/fnut.2021.759507. eCollection 2021. PMID 34901112
- [Background] Crabb DW, Bataller R, Chalasani NP, Kamath PS, Lucey M, Mathurin P, McClain C, McCullough A, Mitchell MC, Morgan TR, Nagy L, Radaeva S, Sanyal A, Shah V, Szabo G; NIAAA Alcoholic Hepatitis Consortia. Standard Definitions and Common Data Elements for Clinical Trials in Patients With Alcoholic Hepatitis: Recommendation From the NIAAA Alcoholic Hepatitis Consortia. Gastroenterology. 2016 Apr;150(4):785-90. doi: 10.1053/j.gastro.2016.02.042. Epub 2016 Feb 24. No abstract available. PMID 26921783
- [Background] Mathurin P, Duchatelle V, Ramond MJ, Degott C, Bedossa P, Erlinger S, Benhamou JP, Chaput JC, Rueff B, Poynard T. Survival and prognostic factors in patients with severe alcoholic hepatitis treated with prednisolone. Gastroenterology. 1996 Jun;110(6):1847-53. doi: 10.1053/gast.1996.v110.pm8964410.
- [Background] Feldman M, FLS and LBJ. Sleisenger and Fordtran's Gastrointestinal and Liver Disease. 2016. 1254 p.
- [Background] Bajaj JS, O'Leary JG, Reddy KR, Wong F, Olson JC, Subramanian RM, Brown G, Noble NA, Thacker LR, Kamath PS; NACSELD. Second infections independently increase mortality in hospitalized patients with cirrhosis: the North American consortium for the study of end-stage liver disease (NACSELD) experience. Hepatology. 2012 Dec;56(6):2328-35. doi: 10.1002/hep.25947. PMID 22806618
- [Background] Daswani R, Kumar A, Anikhindi SA, Sharma P, Singla V, Bansal N, Arora A. Predictors of 90-day mortality in patients with severe alcoholic hepatitis: Experience with 183 patients at a tertiary care center from India. Indian J Gastroenterol. 2018 Mar;37(2):141-152. doi: 10.1007/s12664-018-0842-0. Epub 2018 Apr 28. PMID 29704174
- [Background] Kumar SE, Goel A, Zachariah U, Nair SC, David VG, Varughese S, Gandhi PB, Barpha A, Sharma A, Vijayalekshmi B, Balasubramanian KA, Elias E, Eapen CE. Low Volume Plasma Exchange and Low Dose Steroid Improve Survival in Patients With Alcohol-Related Acute on Chronic Liver Failure and Severe Alcoholic Hepatitis - Preliminary Experience. J Clin Exp Hepatol. 2022 Mar-Apr;12(2):372-378. doi: 10.1016/j.jceh.2021.07.010. Epub 2021 Jul 21. PMID 35535077
- [Background] Plauth M, Cabre E, Riggio O, Assis-Camilo M, Pirlich M, Kondrup J; DGEM (German Society for Nutritional Medicine); Ferenci P, Holm E, Vom Dahl S, Muller MJ, Nolte W; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Liver disease. Clin Nutr. 2006 Apr;25(2):285-94. doi: 10.1016/j.clnu.2006.01.018. Epub 2006 May 16. PMID 16707194
- [Background] https://www.aasld.org/liver-fellow-network/core-series/why-series/why-nutrition-so-important-alcohol-associated-liver, 2022.
- [Background] Arab JP, Diaz LA, Baeza N, Idalsoaga F, Fuentes-Lopez E, Arnold J, Ramirez CA, Morales-Arraez D, Ventura-Cots M, Alvarado-Tapias E, Zhang W, Clark V, Simonetto D, Ahn JC, Buryska S, Mehta TI, Stefanescu H, Horhat A, Bumbu A, Dunn W, Attar B, Agrawal R, Haque ZS, Majeed M, Cabezas J, Garcia-Carrera I, Parker R, Cuyas B, Poca M, Soriano G, Sarin SK, Maiwall R, Jalal PK, Abdulsada S, Higuera-de la Tijera MF, Kulkarni AV, Rao PN, Guerra Salazar P, Skladany L, Bystrianska N, Prado V, Clemente-Sanchez A, Rincon D, Haider T, Chacko KR, Cairo F, de Sousa Coelho M, Romero GA, Pollarsky FD, Restrepo JC, Castro-Sanchez S, Toro LG, Yaquich P, Mendizabal M, Garrido ML, Narvaez A, Bessone F, Marcelo JS, Piombino D, Dirchwolf M, Arancibia JP, Altamirano J, Kim W, Araujo RC, Duarte-Rojo A, Vargas V, Rautou PE, Issoufaly T, Zamarripa F, Torre A, Lucey MR, Mathurin P, Louvet A, Garcia-Tsao G, Gonzalez JA, Verna E, Brown RS, Roblero JP, Abraldes JG, Arrese M, Shah VH, Kamath PS, Singal AK, Bataller R. Identification of optimal therapeutic window for steroid use in severe alcohol-associated hepatitis: A worldwide study. J Hepatol. 2021 Nov;75(5):1026-1033. doi: 10.1016/j.jhep.2021.06.019. Epub 2021 Jun 21. PMID 34166722
- [Background] Van Melkebeke L, Pollentier L, Van der Merwe S, Nevens F, Verbeek J. Letter to the Editor: Survival in placebo-treated patients with severe alcohol-associated hepatitis. Hepatology. 2023 May 1;77(5):E113-E114. doi: 10.1097/HEP.0000000000000336. Epub 2023 Feb 24. No abstract available. PMID 36815362
- [Background] Sidhu S, Goyal O, Gupta A, Kishore H, Gupta A. Corticosteroids and Bovine Colostrum in Treatment of Alcoholic Hepatitis 'In Extremis': A Pilot Study. J Clin Exp Hepatol. 2015 Jun;5:S19-20.
- [Background] Godhia M, Patel N. Colostrum Its Composition, Benefits As A Nutraceutical : A Review. Current Research in Nutrition and Food Science Journal. 2013 Aug 29;1(1):37-47.
- [Background] Dziewiecka H, Buttar HS, Kasperska A, Ostapiuk-Karolczuk J, Domagalska M, Cichon J, Skarpanska-Stejnborn A. A Systematic Review of the Influence of Bovine Colostrum Supplementation on Leaky Gut Syndrome in Athletes: Diagnostic Biomarkers and Future Directions. Nutrients. 2022 Jun 17;14(12):2512. doi: 10.3390/nu14122512. PMID 35745242
- [Background] Halasa M, Maciejewska-Markiewicz D, Baskiewicz-Halasa M, Safranow K, Stachowska E. Post-Delivery Milking Delay Influence on the Effect of Oral Supplementation with Bovine Colostrum as Measured with Intestinal Permeability Test. Medicina (Kaunas). 2020 Sep 24;56(10):495. doi: 10.3390/medicina56100495. PMID 32987647
- [Background] O'Callaghan TF, O'Donovan M, Murphy JP, Sugrue K, Mannion D, McCarthy WP, et al. Evolution of the bovine milk fatty acid profile - From colostrum to milk five days post parturition. Int Dairy J. 2020 May;104:104655
- [Background] Godden S, McMartin S, Feirtag J, Stabel J, Bey R, Goyal S, Metzger L, Fetrow J, Wells S, Chester-Jones H. Heat-treatment of bovine colostrum. II: effects of heating duration on pathogen viability and immunoglobulin G. J Dairy Sci. 2006 Sep;89(9):3476-83. doi: 10.3168/jds.S0022-0302(06)72386-4. PMID 16899682
- [Background] Donahue M, Godden SM, Bey R, Wells S, Oakes JM, Sreevatsan S, Stabel J, Fetrow J. Heat treatment of colostrum on commercial dairy farms decreases colostrum microbial counts while maintaining colostrum immunoglobulin G concentrations. J Dairy Sci. 2012 May;95(5):2697-702. doi: 10.3168/jds.2011-5220. PMID 22541498
- [Background] Bolke E, Orth K, Jehle PM, Schwarz A, Steinbach G, Schleich S, Ulmer C, Storck M, Hannekum A. Enteral application of an immunoglobulin-enriched colostrum milk preparation for reducing endotoxin translocation and acute phase response in patients undergoing coronary bypass surgery--a randomized placebo-controlled pilot trial. Wien Klin Wochenschr. 2002 Nov 30;114(21-22):923-8. PMID 12528325
- [Background] Bolke E, Jehle PM, Hausmann F, Daubler A, Wiedeck H, Steinbach G, Storck M, Orth K. Preoperative oral application of immunoglobulin-enriched colostrum milk and mediator response during abdominal surgery. Shock. 2002 Jan;17(1):9-12. doi: 10.1097/00024382-200201000-00002. PMID 11795674
- [Background] Forrest EH, Gleeson D. Is a liver biopsy necessary in alcoholic hepatitis? J Hepatol. 2012 Jun;56(6):1427-8; author reply 1428-9. doi: 10.1016/j.jhep.2011.12.028. Epub 2012 Feb 3. No abstract available. PMID 22310696
- [Background] Keating M, Lardo O, Hansell M. Alcoholic Hepatitis: Diagnosis and Management. Am Fam Physician. 2022 Apr 1;105(4):412-420. PMID 35426628
- [Derived] Sidhu SS, Dusseja A, Shalimar, Nijhawan S, Kapoor D, Goyal O, Kishore H. A multicenter double-blind, placebo-controlled randomized trial to evaluate the safety and efficacy of bovine colostrum in the treatment of severe alcoholic hepatitis (SAH). Trials. 2023 Aug 11;24(1):515. doi: 10.1186/s13063-023-07505-8. PMID 37568158